CLINICAL TRIAL: NCT00003963
Title: Treatment of B-Cell NHL Relapsing After Transplant With a Rituxan Vinorelbine Combination
Brief Title: Chemotherapy and Monoclonal Antibody Therapy in Treating Patients With B-cell Non-Hodgkin's Lymphoma That Has Relapsed Following Peripheral Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Christos Emmanouilides, MD / Principal Investigator, UCLA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067163; UCLA-9903029; NCI-G99-1545
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-07

CONDITIONS: Lymphoma
Keywords: Waldenstrom macroglobulinemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vinorelbine and Rituxan (Experimental): Week 1-4: Rituxan is given at 375 mg/m2 weekly x4. Vinorelbine (25mg/m2) given 1 week after the first rituxan dose and immediately after the second rituxan dose.
  Week 5-8: Rituxan given every 2 weeks. Vinorelbine given weekly x3, with one week off.
  Week 9-12: Schedule same as week 5-8. Week 13 and following: If subject doesn't have disease progression, they may continue on Vinorelbine until progression or until clinically indicated.
  Interventions: Biological: rituximab; Drug: vinorelbine ditartrate

INTERVENTIONS:
Biological: rituximab — Week 1-4: Rituxan is given at 375 mg/m2 weekly x4. Week 5-8: Rituxan given every 2 weeks. Week 9-12: Schedule same as week 5-8.
  Other Names: Rituxan
Drug: vinorelbine ditartrate — Week 1-4: Vinorelbine (25mg/m2) given 1 week after the first rituxan dose and immediately after the second rituxan dose.
  Week 5-8: Vinorelbine given weekly x3, with one week off. Week 9-12: Schedule same as week 5-8. Week 13 and following: If subject doesn't have disease progression, they may continue on Vinorelbine until progression or until clinically indicated.
  Other Names: Vinorelbine

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining monoclonal antibody therapy with chemotherapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of the monoclonal antibody rituximab plus chemotherapy with vinorelbine in treating patients with B-cell non-Hodgkin's lymphoma that has relapsed following autologous peripheral stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the tolerability and toxicity of rituximab combined with vinorelbine in patients with relapsed non-Hodgkin's lymphoma following autologous peripheral blood stem cell transplantation.
* Assess the response rate and duration of response to this regimen in these patients.

OUTLINE: Patients receive rituximab IV weekly on weeks 1-4, 6, 8, 10, and 12 and vinorelbine IV on weeks 2-4, 6-8, and 10-12. Patients who achieve partial response may continue on vinorelbine from week 14 until disease progression.

Patients are followed until disease progression.

PROJECTED ACCRUAL: A total of 18-25 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with B-cell Lymphoma, relapsing after high dose chemotherapy and autologous stem cell transplantation or allogeneneic stem cell or bone marrow transplant
* Age > 18 years old
* Adequate hematologic function, as manifested by ANC > 1000/mm3 and platelet count > 40,000/mm3
* PS WHO: < 3

Exclusion Criteria:

* Patients with serum creatinine > 2 mg%, transaminases (ALT, AST) > 3 times upper normal value, direct bilirubin > 2 mg%, unless they result from tumor involvement
* Pregnant or lactating females
* History of myelodysplastic syndrome
* Uncontrolled CNS disease
* Active serious infection
* History of refractoriness to vinorelbine. However, prior treatment with rituxan is not an exclusion (synergy may still occur)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 1999-05; Primary Completion 2003-09 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Tolerability and toxicity | 13 weeks
  To define the tolerability and toxicity of a combination regimen of rituxan combined with vinorelbine for the treatment of B-cell NHL, relapsing after autologous stem cell transplantation.

SECONDARY OUTCOMES:
Response rate | 13 weeks
  To preliminarily assess the response rates to such a regimen; to assess duration of response.

CONTACTS AND LOCATIONS:
Overall Officials: Christos E. Emmanouilides, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States